CLINICAL TRIAL: NCT05444322
Title: A Study of RD14-01 in Patients With Relapsed or Refractory B Cell Non-Hodgkin Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: He Huang (Other)
Responsible Party: Sponsor-Investigator, He Huang, Clinical Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD14-01
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Mantle Cell Lymphoma; Diffuse Large B-cell Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD14-01 cell infusion (Experimental): Infused i.v. in a single dose
  Interventions: Drug: RD14-01 cell infusion

INTERVENTIONS:
Drug: RD14-01 cell infusion — Autologous CAR T cells

SUMMARY:
This study is designed to explore the safety and tolerability of RD14-01 for patients with relapsed and/or refractory B-cell non-Hodgkin lymphoma. And to evaluate the efficacy and pharmacokinetics of RD14-01 in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years.
2. Diagnosis of r/r MCL, DLBCL, or FL (Grade 1, 2 and 3a).
3. ECOG: 0-1.
4. Life expectancy greater than 3 months.
5. Cardiac left ventricle ejection fraction ≥50%.
6. Informed consent explained to, understood by and signed by the patient/guardian. Patient/guardian is given a copy of informed consent.

Exclusion Criteria:

1. Pregnant or lactating.
2. Hepatitis B surface antigen (HBsAg) or hepatitis B e-antigen (HBeAg) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal range; hepatitis C virus (HCV) antibody positive; human immunodeficiency virus (HIV) antibody positive; syphilis antibody positive; cytomegalovirus (CMV) DNA positive; Epstein-Barr virus (EBV) DNA positive.
3. Central nervous system (CNS) metastases.
4. Participated in other clinical studies within 4 weeks prior to screening.
5. History of alcoholism, drug abuse or mental illness.
6. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 2 years
  DLT
Maximum tolerable dose | Up to 2 years
  MTD

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No